CLINICAL TRIAL: NCT06839703
Title: International Open-label Phase I Dose Escalation Study of Dinutuximab Beta in Combination With Vincristine/Doxorubicin/Cyclophosphamide and Ifosfamide/Etoposide in Pediatric, Adolescent, and Adult Patients With GD2-positive Ewing Sarcoma
Brief Title: International Phase I Trial of Dinutuximab Beta With VDC/IE in GD2-Positive Ewing Sarkoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Dr. Dirk Reinhardt (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dirk Reinhardt, Por. Dr. Dirk Reinhardt, German Society for Pediatric Oncology and Hematology GPOH gGmbH
Organization: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CESS-GD2
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: High-risk GD2-Positive Ewing Sarcoma
Keywords: Biomarker; GD2 expression; targeted therapy; high-risk Ewing Sarcoma
MeSH Terms: interventions — dinutuximab

STUDY DESIGN:
Intervention Model Description: This is a multi-center, phase 1, open-label, dose escalation study enrolling high-risk Ewing sarcoma patients that have been tested with GD2-positivity in a classical 3+3 design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dinutuximab beta added to standard chemotherapy (Experimental): Dinutuximab beta is added in different dosages to the standard chemotherapy
  Interventions: Drug: Dinutuximab beta

INTERVENTIONS:
Drug: Dinutuximab beta — Dinutuximab beta is added in different dosages to the standard chemotherapy

SUMMARY:
The goal of the study is to investigate the feasibility, toxicity, and biological activity of the treatment with dinutuximab beta in combination with standard chemotherapy in EWS to give high-risk patients with a GD2 positiv pumor a benefit in treatment. Within the study is tested with three different dosages in a 3+3 design with three pre-defined dose levels.

DETAILED DESCRIPTION:
Immunotherapeutic approaches have emerged as an effective therapeutic approach in cancer. We will investigate the cell-surface ganglioside GD2 as a target since it is expressed on the cell surface of Ewing Sarcoma cells and clinical trials support the safety and efficacy of anti-GD2 antibodies in pediatric solid cancers.

Dinutuximab beta is a chimeric antibody that targets the disialoganglioside GD2. GD2 is expressed on a number of solid malignancies and was clinically investigated in pediatric patients with neuroblastoma. Expression in normal tissues is restricted to cerebellar neurons, skin melanocytes and peripheral pain fibers. Due to this expression pattern, anti-GD2 antibodies have been studied as targeted immunotherapy for neuroblastoma. With the results of these clinical trials, combination therapies with dinutuximab beta became a standard component of high-risk neuroblastoma therapy. GD2 expression is found in several EWS samples with variable expression-levels, and it is expected that anti-GD2 treatment is best suited as biomarker-driven approach.

The administration of vincristine, doxorubicin, cyclophosphamide, ifosfamide and etoposide (VDC/IE) has been shown to be an effective systemic therapy and is therefore currently part of the standard treatment in Ewing Sarcoma. The international newest standard induction chemotherapy in the standard- and high-risk group consists of alternating VDC/IE. High-risk patients with a GD2 positive tumor could benefit from an addition of dinutuximab beta to the standard chemotherapy with VDC/IE.

The rationale for this trial is to investigate the feasibility, toxicity, and biological activity of dinutuximab beta in combination with standard chemotherapy in EWS.

This is a multi-center, phase 1, open-label, dose escalation study enrolling high-risk Ewing sarcoma patients that have been tested with GD2-positivity in a classical 3+3 design.

The decision to initiate treatment with 50% of the approved dosage for neuroblastoma in this dose-escalation study is grounded in both scientific literature and safety considerations. Starting at a lower dosage allows for the careful monitoring of patient response and minimizes the risk of adverse effects, particularly in a dose-sensitive adult population.

A risk assessment further supports this approach, indicating that starting at 50% of the approved neuroblastoma dose provides a safe baseline from which to escalate. The assessment outlines that a stepwise increase to 75% and subsequently to 100% of the approved dose allows for the identification of any dose-limiting toxicities (DLTs) in a controlled manner, thus optimizing patient safety.

The choice of 100 mg/m2 as the maximum dosage per cycle, equivalent to the dosage used in standard neuroblastoma treatment, is justified by its established efficacy and safety profile in this specific indication. The literature supports that doses up to 100 mg/m2 per cycle are well-tolerated in the majority of patients, with the therapeutic benefits outweighing the risks when administered within a carefully monitored clinical framework.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed Ewing Sarcoma (m/f/d) or so-called Ewing-like sarcoma (i.e. translocation-positive small blue round cell sarcoma other than Rhabdomyosarcoma) of bone and / or soft tissue with evidence of EWS translocation by fluorescence in situ hybridization (FISH), real-time polymerase chain reaction (RT-PCR), or next-generation sequencing (NGS) assay
2. High risk stratification (metastatic disease)
3. Centrally confirmed GD2-positive tumor (biopsy of original and/or residual tumor or liquid biopsy in peripheral blood)
4. Availability of fresh frozen tumor tissue for central GD2-detection
5. Age ≥12 months
6. Start of first line treatment according to standard induction treatment (Cycle 1-4: VDC - IE - VDC - IE)
7. Wash-out phase with a minimum of 14 days after the last the dose of the last chemotherapy
8. Lansky (<16 years) Performance Score ≥70% or ECOG (≥16 years) ≤ 2
9. Adequate bone marrow function as evidenced by meeting all the following requirements:

   1. White blood cell count > 2000/μl
   2. ANC ≥1000 cells/μL (G-CSF allowed)
   3. Platelet count 75,000 cells/μL without the use of platelet transfusion within the last 2 days
   4. Hemoglobin ≥9 g/dL without the use of red blood cell transfusion within the last 2 days
10. Adequate hepatic function as evidenced by meeting all the following requirements:

    1. Serum total bilirubin ≤1.5 x upper limit of normal (ULN)
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x ULN
11. Adequate cardiac function: confirmed by echocardiography with a left ventricular ejection fraction (LVEF) of ≥ 50%
12. Adequate renal function: creatinine clearance or glomerular filtration rate (GFR) > 60 mL/min/1.73 m2
13. No known active HIV, HBV, or HCV infection
14. No severe neurological impairment, particularly no motor or sensory deficits, except for neurological deficits caused by Ewing sarcoma
15. Female patients of childbearing potential must present with a negative serum pregnancy test and agree to employ adequate birth control measures for the duration of the study and until 3 months after the end of treatment. Female patients who are lactating must agree to stop breast-feeding from the start of study treatment until 1 month after the end of treatment.
16. Patient or their legal representative is willing and able to comply with the requirements of the study protocol

Exclusion Criteria:

1. Relapsed or refractory Disease state
2. Patients with hypersensitivity against at least 1 component of the investigational medicinal product
3. Significant illnesses and/or any of the following:

   * significant psychiatric disabilities or uncontrolled seizure disorders
   * active uncontrolled peptic ulcer disease
   * clinically significant neurologic deficit or objective peripheral neuropathy
   * clinically significant, symptomatic fluid in a third space
4. Active and uncontrolled CNS metastases (indicated by clinical symptoms, cerebral edema, corticosteroid and/or anticonvulsant requirement, or progressive disease); for controlled CNS metastases, patient should have been off corticosteroids for at least 28 days without overt evidence of significant neurological deficits prior to enrollment
5. Significant cardiac conduction abnormalities, including known familial prolonged QT syndrome, or screening QTc >480 msec
6. Active, uncontrolled infection or an unexplained fever >38.5°C which in the Investigator's opinion might compromise the patient's participation in the study or affect the study outcome
7. Chronic Grade ≥2 diarrhea
8. Diagnosis of any malignancy other than the disease under study
9. Any other medical or social condition deemed by the Investigator to be likely to interfere with a patient's ability to cooperate and participate in the study or interfere with the interpretation of the results.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
GD2 Positivity | after initial diagnosis and before study enrolment
  local assessment for GD2 positivity

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06839703/Prot_000.pdf